CLINICAL TRIAL: NCT05385822
Title: Pelvic Floor Muscle Training in the Treatment of Erectile Dysfunction: A Randomized, Controlled Trial
Brief Title: Pelvic Floor Muscle Training in the Treatment of Erectile Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Emil Durukan, Medical Doctor, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRE-Train Project
Record Dates: First submitted 2022-05-04; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Erectile Dysfunction
Keywords: Pelvic Floor Muscle; Erectile Dysfunction; Sexual Dysfunction; Impotence; Kegel Exercise; Training
MeSH Terms: conditions — Erectile Dysfunction; Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: Men who meet all inclusion criteria will be randomized 1:1 for either pelvic floor training or control. Stratified randomization with correction for IIEF-EF category is used (mild 17-25, moderate 11-16, severe 0-10)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will not recieve any training in the trial period but will have to answer the same questionnaires on erectile function (IIEF-EF) and international prostate symptom score (IPSS).
- Pelvic Floor Muscle Training (Experimental): Participants who are randomized to pelvic floor training will then undergo instruction in the anatomy, function and training of the pelvic floor muscles.
  Interventions: Behavioral: Pelvic Floor Muscle Training

INTERVENTIONS:
Behavioral: Pelvic Floor Muscle Training — * Isolated, quite light tension in the pelvic floor 10 times, where the tension is released immediately
  * Constant tension for 30 seconds twice, with a 30-second pause
  * Total relaxation for 1 minute They must perform these exercises once a day during the trial period of 3 months
  Arms: Pelvic Floor Muscle Training

SUMMARY:
Erectile dysfunction affects about 40% of all men above the age of 40 and the prevalence increases with increasing age. It is not possible to cure the condition as current forms of treatment are aimed solely at improving symptoms. Treatment options today include medications, injection therapy, and vacuum pumps, among others. However, pelvic floor muscle training is a natural, inexpensive, and non-invasive form of treatment that is used to a limited extent.

Theoretically, a strengthening of the pelvic floor muscles can help increase the intracavernous pressure and thereby the hardness of the erection. Furthermore, tense pelvic floor muscles can help compress pelvic veins and reduce blood flow away from the penis which prolongs the erection. Finally, it is possible that pelvic floor muscle training can contribute to an increased blood supply to the pelvic floor and the penis which will have positive effects in relation to both the integrity of the penile tissue and the physiological erection mechanism itself.

This study aims to investigate the effect of pelvic floor muscle training in men with erectile dysfunction.

The study hypothesis is that pelvic floor training can provide a clinically significant improvement in the erection function at individual patient level

ELIGIBILITY:
Inclusion Criteria:

* Erectile Dysfunction for more than 6 months
* IIEF-EF score < 25
* In a stable heterosexual relationship in minimum of 3 months (since all questionnaires are only validated for heterosexuals)

Exclusion Criteria:

* Known psychiatric, neurological, and/or endocrine disorders (including hypogonadism with total testosterone <12 nmol / l)
* Traumatic nerve damage
* Diabetes
* Previous surgery or radiotherapy in the pelvic region
* Nerve disorders that prevent nerve connection to the pelvic floor muscles
* Severe heart disease in the form of unstable angina, NYHA class > II heart failure, uncontrolled arrhythmia or severe symptomatic and/or severe valvular disease
* Use of anti-androgen drugs Peyronie's disease and/or previous cases of priapism
* Alcohol overconsumption (more than 21 items per week)

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Clinically significant improvements in erectile function | 1 month after first pelvic floor muscle training session
  The proportion of patients who achieve clinically significant improvements in the erectile function (EF) domain of the International Index of Erectile Function (IIEF) after 3 months of pelvic floor training or observation in an intention-to-treat analysis (assessed 1 month after the last training session). This is defined according to Rosen et al. (mild ED: 2 points; moderate ED: 5 points; severe ED: 7 points)
Clinically significant improvements in erectile function | 4 months after first pelvic floor muscle training session
  The proportion of patients who achieve clinically significant improvements in the erectile function (EF) domain of the International Index of Erectile Function (IIEF) after 3 months of pelvic floor training or observation in an intention-to-treat analysis (assessed 1 month after the last training session). This is defined according to Rosen et al. (mild ED: 2 points; moderate ED: 5 points; severe ED: 7 points)
Clinically significant improvements in erectile function | 6 months after first pelvic floor muscle training session
  The proportion of patients who achieve clinically significant improvements in the erectile function (EF) domain of the International Index of Erectile Function (IIEF) after 3 months of pelvic floor training or observation in an intention-to-treat analysis (assessed 1 month after the last training session). This is defined according to Rosen et al. (mild ED: 2 points; moderate ED: 5 points; severe ED: 7 points)
Clinically significant improvements in erectile function | 12 months after first pelvic floor muscle training session
  The proportion of patients who achieve clinically significant improvements in the erectile function (EF) domain of the International Index of Erectile Function (IIEF) after 3 months of pelvic floor training or observation in an intention-to-treat analysis (assessed 1 month after the last training session). This is defined according to Rosen et al. (mild ED: 2 points; moderate ED: 5 points; severe ED: 7 points)

SECONDARY OUTCOMES:
Changes in the International Index of Erectile Function questionnaire category; orgasmic function. Items 9-10. Score range: 0-5. Maximum score: 10. | 1 month after first pelvic floor muscle training session
  Low score points represent a reduced orgasmic function whereas high score points represent a better/improved orgasmic function. The scores will be calculated and compared between groups as continuous variables.
Changes in the International Index of Erectile Function questionnaire category; orgasmic function. Items 9-10. Score range: 0-5. Maximum score: 10. | 4 months after first pelvic floor muscle training session
  Low score points represent a reduced orgasmic function whereas high score points represent a better/improved orgasmic function. The scores will be calculated and compared between groups as continuous variables.
Changes in the International Index of Erectile Function questionnaire category; orgasmic function. Items 9-10. Score range: 0-5. Maximum score: 10. | 6 months after first pelvic floor muscle training session
  Low score points represent a reduced orgasmic function whereas high score points represent a better/improved orgasmic function. The scores will be calculated and compared between groups as continuous variables.
Changes in the International Index of Erectile Function questionnaire category; orgasmic function. Items 9-10. Score range: 0-5. Maximum score: 10. | 12 months after first pelvic floor muscle training session
  Low score points represent a reduced orgasmic function whereas high score points represent a better/improved orgasmic function. The scores will be calculated and compared between groups as continuous variables.
Changes in the International Index of Erectile Function questionnaire category; sexual desire. Items 11-12. Score range: 1-5. Maximum score: 10. | 1 month after first pelvic floor muscle training session
  Low score points represent a reduced sexual desire whereas high score points represent a high sexual desire. The scores will be calculated and compared between groups as continuous variables.
Changes in the International Index of Erectile Function questionnaire category; sexual desire. Items 11-12. Score range: 1-5. Maximum score: 10. | 4 months after first pelvic floor muscle training session
  Low score points represent a reduced sexual desire whereas high score points represent a high sexual desire. The scores will be calculated and compared between groups as continuous variables.
Changes in the International Index of Erectile Function questionnaire category; sexual desire. Items 11-12. Score range: 1-5. Maximum score: 10. | 6 months after first pelvic floor muscle training session
  Low score points represent a reduced sexual desire whereas high score points represent a high sexual desire. The scores will be calculated and compared between groups as continuous variables.
Changes in the International Index of Erectile Function questionnaire category; sexual desire. Items 11-12. Score range: 1-5. Maximum score: 10. | 12 months after first pelvic floor muscle training session
  Low score points represent a reduced sexual desire whereas high score points represent a high sexual desire. The scores will be calculated and compared between groups as continuous variables.
Changes in the International Index of Erectile Function questionnaire category; intercourse satisfaction. Items 6-8. Score range: 0-5. Maximum score: 15. | 1 month after first pelvic floor muscle training session
  Low score points represent a reduced intercourse satisfaction whereas high score points represent high intercourse satisfaction. The scores will be calculated and compared between groups as continuous variables.
Changes in the International Index of Erectile Function questionnaire category; intercourse satisfaction. Items 6-8. Score range: 0-5. Maximum score: 15. | 4 months after first pelvic floor muscle training session
  Low score points represent a reduced intercourse satisfaction whereas high score points represent high intercourse satisfaction. The scores will be calculated and compared between groups as continuous variables.
Changes in the International Index of Erectile Function questionnaire category; intercourse satisfaction. Items 6-8. Score range: 0-5. Maximum score: 15. | 6 months after first pelvic floor muscle training session
  Low score points represent a reduced intercourse satisfaction whereas high score points represent high intercourse satisfaction. The scores will be calculated and compared between groups as continuous variables.
Changes in the International Index of Erectile Function questionnaire category; intercourse satisfaction. Items 6-8. Score range: 0-5. Maximum score: 15. | 12 months after first pelvic floor muscle training session
  Low score points represent a reduced intercourse satisfaction whereas high score points represent high intercourse satisfaction. The scores will be calculated and compared between groups as continuous variables.
Changes in the International Index of Erectile Function questionnaire category; overall satisfaction. Items 13-14. Score range: 1-5. Maximum score: 10. | 1 month after first pelvic floor muscle training session
  Low score points represent a reduced overall satisfaction whereas high score points represent high overall satisfaction. The scores will be calculated and compared between groups as continuous variables.
Changes in the International Index of Erectile Function questionnaire category; overall satisfaction. Items 13-14. Score range: 1-5. Maximum score: 10. | 4 months after first pelvic floor muscle training session
  Low score points represent a reduced overall satisfaction whereas high score points represent high overall satisfaction. The scores will be calculated and compared between groups as continuous variables.
Changes in the International Index of Erectile Function questionnaire category; overall satisfaction. Items 13-14. Score range: 1-5. Maximum score: 10. | 6 months after first pelvic floor muscle training session
  Low score points represent a reduced overall satisfaction whereas high score points represent high overall satisfaction. The scores will be calculated and compared between groups as continuous variables.
Changes in the International Index of Erectile Function questionnaire category; overall satisfaction. Items 13-14. Score range: 1-5. Maximum score: 10. | 12 months after first pelvic floor muscle training session
  Low score points represent a reduced overall satisfaction whereas high score points represent high overall satisfaction. The scores will be calculated and compared between groups as continuous variables.
Participant satisfaction | 4 months after first pelvic floor muscle training
  Subjective participant satisfaction assessed using a modified version of the patient version of the Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) questionnaire after treatment. This analysis will be performed as an intention-to-treat analysis without correction for missing data. Each EDITS item is scored from 0 to 4, with higher scores indicating greater treatment satisfaction. The mean EDITS questionnaire score is multiplied by 25, yielding a standardized EDITS index of treatment satisfaction score, ranging from 0 (low satisfaction) to 100 (extremely high satisfaction).
Changes in the International Prostate Symptom Score | 1 month after first pelvic floor muscle training session
  Changes in the International Prostate Symptom Score will be assessed from all the participants. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Changes in the International Prostate Symptom Score | 6 months after first pelvic floor muscle training session
  Changes in the International Prostate Symptom Score will be assessed from all the participants. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Changes in the International Prostate Symptom Score | 12 months after first pelvic floor muscle training session
  Changes in the International Prostate Symptom Score will be assessed from all the participants. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Urological Research Unit, Herlev, Capital Region, Denmark